CLINICAL TRIAL: NCT00955578
Title: Identification of the Genetic Mutation Responsible for Segmental Dysplastic Nevi
Brief Title: Genetic Identification (ID) of Segmental Dysplastic Nevi
Status: Withdrawn | Type: Observational
Why Stopped: Study was not submitted or reviewed by the NSH REB, reason unknown
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: SDN-001
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2009-09

CONDITIONS: Segmental Dysplastic Nevi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The participant will be involved in the study for the length of time required to obtain 5 to 6 skin biopsiesThe laboratory testing that will be performed includes a genetic analysis of the tissue obtained from biopsy. The genetic analysis will take place in the genetics lab of Dr. Hensin Tsao, Massachusetts General Hospital, Bartlett 622, 48 Blossom Street, Boston MA, 02114.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Segmental Dysplastic Nevi: One patient who has been diagnosed with SDN and has had previous biopsies in the past, comparing to current biopsies
  Interventions: Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Punch Biopsy — 5-6 punch biopsies of affected areas

SUMMARY:
The investigators' goal is to identify the mutation in the gene that is responsible for the development of segmental dysplastic nevi. To identify the gene the investigators may use a candidate gene approach (i.e. sequence specific genes that are thought to be involved: NRAS, BRAF, etc) or a genome-wide approach trying to implicate regions in the genome (Loss-of-heterozygosity or copy number changes on comparative genomic hybridization).

DETAILED DESCRIPTION:
Dysplastic (atypical) melanocytic (DMN) nevi have been identified as being potential precursors of melanoma and markers for patients at risk of developing primary melanoma1. In addition, having an increased number of nevi is associated with increased risk1. DMN are present in 2-5% of white adults in the U.S. population and international studies have documented up to 18% prevalence2. These lesions may be present in at least 17% of white adults with melanoma and 20-50% of melanomas may arise in nevi and atypical nevi2. The exact gene(s) involved in the development of nevi have yet to be elucidated.

Segmental dysplastic nevi are nevi that are restricted to one area of the body3. This condition is much rarer than the occurrence of dysplastic nevi, but nonetheless, may involve the same genetic mutation. The pattern of distribution in SDN is thought to result from mosaicism, i.e. the part of the body that expresses the dysplastic nevi has a mutation in a gene, however, the rest of the body does not contain this same mutation. Other mosaic disorders that have been studied in greater detail than SDN have been shown to be caused by a single gene mutation4. It appears that SDN is no different and that it too is caused by a mutation in a single gene, however, this gene is not yet known.

In this study we will perform a genetic analysis of tissue from a patient known to have SDN. With the information we gather from this analysis, we may be able to find the gene responsible for the development of dysplastic nevi.

Primary Research Objective:

To investigate the genetic mutation involved in the development of dysplastic nevi by examining a patient with SDN.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a positive history of segmental dysplastic nevi

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One patient who is already known to the principal investigator
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12; Study Completion 2010-03

CONTACTS AND LOCATIONS:
Overall Officials: Richard GB Langley, MD, FRCPC, Principal Investigator — Capital Health/Dalhousie University
Locations (1):
- Capital Heatlh, Halifax, Nova Scotia, Canada